CLINICAL TRIAL: NCT04184726
Title: Mindfulness Based Cognitive Therapy Modified for Visual Symptoms: MBCT-vision
Brief Title: Mindfulness Based Cognitive Therapy Modified for Visual Symptoms (MBCT-vision)
Acronym: MBCT-vision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 266101
Record Dates: First submitted 2019-11-26; First posted 2019-12-04 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2022-01

CONDITIONS: Visual Snow Syndrome; Trailing Phenomenon; Photophobia; Visual Aura
Keywords: Mindfulness; Mindfulness Based Cognitive Therapy
MeSH Terms: conditions — visual snow syndrome; Photophobia; Epilepsy, Partial, Sensory | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: MBCT-vision intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MBCT-vision (Experimental): 8 x once weekly group sessions, and home practice between sessions
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy — mindfulness and cognitive behavioural therapy techniques taught in group sessions meeting once weekly for 8 weeks, and home practice between sessions.
  Other Names: MBCT

SUMMARY:
This is a research study on Mindfulness-Based Cognitive Therapy for visual symptoms (MBCT-vision), to treat patients with debilitating symptoms of visual snow (VS) and is associated visual symptoms, severe light sensitivity (i.e. photophobia) and migrainous visual aura.

Participants will receive an intervention of an 8-week MBCT course modified for visual symptoms, which will involve 8 weeks of once weekly group sessions and home practice between sessions.

DETAILED DESCRIPTION:
This is a research study on Mindfulness-Based Cognitive Therapy for visual symptoms (MBCT-vision), to treat patients with debilitating symptoms of visual snow (VS) and its associated visual symptoms, severe light sensitivity (i.e. photophobia) and migrainous visual aura.

VS is a condition of persistent flickering dots, like that of an out-of-focus analog television screen, affecting the whole visual field. There can be associated visual symptoms such as after-images, and trailing of images. No clinical trials for treatment have been done for VS. Instead, treatment data comes from patient case reports.

Photophobia describes discomfort or pain to light stimulation. Causes include eye surface issues, migraine, or of an unknown trigger, and can be persistent despite optimum management of underlying causes.

Patients with migrainous visual aura may have troublesome visual disturbances despite optimum migraine treatment.

Previous studies have shown that dysfunction in brain pathways contribute to the above conditions.

Mindfulness-Based Cognitive Therapy is a treatment that combines evidence-based approaches of Mindfulness-Based Stress Reduction and Cognitive Behavioural Therapy (CBT). MBCT is an established 8-week programme designed to develop skills of mindfulness and CBT strategies in individuals, through weekly small-group sessions and structured daily practice between sessions.

Studies on MBCT and mindfulness-based interventions have shown improvements in psychological resilience; physical health including immune function; and neural changes associated with psychological wellbeing.

The investigators propose that MBCT, modified to incorporate aspects relevant to persistent and distressing visual symptoms (MBCT-vision), can improve these debilitating symptoms by modifying dysfunctional neural pathways and equip patients with skills that promote psychological resilience and improve coping with residual symptoms.

For this study, the investigators will assess the use of MBCT-vision in patients with visual snow or associated visual symptoms, migrainous visual aura or photophobia. This will be the first study of a mindfulness-based intervention in this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with visual snow or associated visual symptoms; photophobia for at least 3 months
* Patients with migrainous visual aura occurring >4 episodes a month for at least 3 months

Exclusion Criteria:

* Patient with a current severe depressive or psychotic episode
* Patient with severe difficulties in emotional regulation
* Patient unable to provide informed consent for participation
* Patient with insufficient understanding of spoken English (due to need to participate in group discussions)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
change in severity of visual symptoms | week 9 and 20
  change in severity of visual symptoms pre- and post-intervention, comparing scores on Likert scale, ranging from 0/10 (no symptoms) to 10/10 (extremely severe symptoms)

SECONDARY OUTCOMES:
change in World Health Organisation (WHO) wellbeing index scores | week 9 and 20
  change in WHO wellbeing index, comparing pre- and post- intervention scores. WHO wellbeing index range from 0-25, with higher scores representing increased wellbeing.
change in Clinical Outcomes in Routine Evaluation (CORE-10) scores | week 9 and 20
  change in CORE-10 scores, comparing pre- and post- intervention. CORE-10 scores range from 0-40 with higher scores indicating more distress.
change in Five-Facet Mindfulness Questionnaire (FFMQ) scores | week 9 and 20
  change in Five-Facet Mindfulness Questionnaire scores, comparing pre- and post- intervention. FFMQ scores range from 39-195 where higher scores represent more mindfulness
compliance (session attendance and completion of daily practice) | week 9
  participant compliance from attendance record for MBCT-vision weekly sessions and self-report compliance with daily home practice
qualitative assessment of MBCT-vision | week 9
  participant feedback on the design of MBCT-vision via structured qualitative interview
functional MRI | week 20
  changes to functional MRI comparing baseline to week 20 - this has been added for participants recruited in the second and third cohort

CONTACTS AND LOCATIONS:
Overall Officials: Sui H Wong, MD, Principal Investigator — Guys & St Thomas'
Locations (1):
- Guys & St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong SH, Pontillo G, Kanber B, Prados F, Wingrove J, Yiannakas M, Davagnanam I, Gandini Wheeler-Kingshott CAM, Toosy AT. Visual Snow Syndrome Improves With Modulation of Resting-State Functional MRI Connectivity After Mindfulness-Based Cognitive Therapy: An Open-Label Feasibility Study. J Neuroophthalmol. 2024 Mar 1;44(1):112-118. doi: 10.1097/WNO.0000000000002013. Epub 2023 Nov 15. PMID 37967050